CLINICAL TRIAL: NCT06666777
Title: Speech Therapy and Parenting for Early Socio-communicative Skills in Children With Neurodevelopmental Disabilities
Brief Title: Speech Therapy and Parenting for Early Socio-communicAtive sKills
Acronym: SPEAK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Collaborators: Associazione La Nostra Famiglia, Como, Italy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1109
Record Dates: First submitted 2024-10-08; First posted 2024-10-31 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Neurological Impairments; Genetic Syndrome; Neurodevelopmental Disability; Developmental Delays; Language Development Disorders
Keywords: Socio-communicative skills; early intervention; Speech therapy; Parenting; Parental support; Intersubjectivity; Neurodevelopmental disabilities
MeSH Terms: conditions — Genetic Diseases, Inborn; Language Development Disorders; Communication Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Psychologists administering the Bayley-III Socio-Emotional Questionnaire and ESB Battery, as well as evaluating parenting behavior using the PICCOLO, will be blinded to each participant's group assignment. However, due to the nature of the assessments and treatment, the therapists conducting OPISCoS cannot be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm involving parents (Experimental): Subjects assigned to this arm will receive the intervention focused on intersubjective prelinguistic and socio-communicative skills. A parent is required to participate in all sessions.
  Interventions: Behavioral: Intervention focused on intersubjective prelinguistic and socio-communicative skills
- Standard speech therapy (Active Comparator): Participants in this group will receive standard speech therapy. Parental involvement will only occur if strictly necessary.
  Interventions: Behavioral: Standard speech therapy intervention

INTERVENTIONS:
Behavioral: Intervention focused on intersubjective prelinguistic and socio-communicative skills — The intervention consists of 8 45-minute, weekly sessions over two months. These sessions may take place in various settings, such as free play, snack time, or structured activities. The speech therapist will use these settings to help parents observe intersubjective and social-communicative behaviors, providing guidance and strategies to support them.
  The following topics will be addressed: Early dyadic interaction; First signals of comprehension; Communicative intentionality; Gestures; Attention; Verbal and motor routine; Lexical and syntactic comprehension; Socio-conversational skills.
  These topics are not structured into rigid levels for each session. Instead, several topics may be addressed within the same session and revisited across multiple sessions. This flexibility allows the speech therapist to adapt the intervention based on observations, interactions with the child, and discussions with the parent. Parents in the IG arm will receive a bespoke designed booklet containing
  Other Names: SPEAK
  Arms: Experimental arm involving parents
Behavioral: Standard speech therapy intervention — The standard speech therapy intervention, as typically conducted in rehabilitation centers, consists of 8 weekly sessions, each lasting 45 minutes, over a two-month period (same as the experimental intervention). During these sessions, the therapist may provide various stimulations aimed at enhancing the child's vocalization, verbal comprehension, and speech production. While the therapist may offer guidance to parents on how to continue these stimulations in daily routines, they will not be directly involved in the sessions unless strictly necessary.
  Arms: Standard speech therapy

SUMMARY:
Every year, millions of children are diagnosed with neurodevelopmental disabilities. This term covers a wide range of conditions, from genetic syndromes to brain injuries such as cerebral palsy. Children with neurodevelopmental disabilities often struggle in multiple areas, including language development. While standard speech therapy mainly focuses on understanding and producing words, these children may also have difficulties with the social and communicative skills needed for language. The parent-child relationship is especially important for helping kids develop in their early years.

This clinical trial aims to find out if an intervention focused on early social and communication skills, and involving parents, can help children with neurodevelopmental disabilities. The study includes children aged 6 months to 5 years. It seeks to answer two key questions:

* Does this intervention improve social and communication skills better than standard speech therapy?
* Does this intervention affect how parents interact with their child?

To find the answers, the study will compare two groups: one group will get the parent-involved intervention that focuses on early communication skills, while the other group will get standard speech therapy.

In the first intervention, therapists will guide parents in observing and supporting their child's social and communication behaviors during various activities like playtime and snack time. In contrast, the standard speech therapy will focus on traditional goals, such as improving the child's ability to vocalize, understand, and use words, without involving parents.

Both interventions will follow the same schedule-eight weekly sessions, each lasting 45 minutes, over two months.

Before and after the interventions, the children and parents will:

* Have an assessment of the child's language, social, and communication development.
* Participate in a 10-minute video recording of parent-child playtime, which will be used to study parenting behavior.

DETAILED DESCRIPTION:
Background: Every year millions of children receive a diagnosis of neurodevelopmental disability (NDD), with a systematic report documenting a prevalence rate estimated in 13.3% of children younger than 5 years in 195 countries. The term neurodevelopmental disability includes diverse clinical conditions ranging from congenital disorders, such as genetic syndromes, to acquired brain damage, such as cerebral palsy. From birth, children with NDD often show difficulties in different developmental domains. For instance, these children may exhibit atypical interactive and attentional skills, they may use less vocal and affective signals and also display difficulties in emotional-behavioral regulation. Such altered interactional and behavioral patterns affect the development of primary intersubjectivity, which refers to the attentional and emotional coordination between parent and child during face-to-face exchanges. Additionally, these challenges can hinder the development of secondary intersubjectivity, where both the parent and child focus their attention on a shared object in the environment. These forms of intersubjectivity are crucial for the emergence of verbal communication. Nonetheless, these abilities are not easily measured by conventional assessments during early childhood, which may result in delayed identification and promotion of early intervention. Assessing and addressing these early socio-communicative difficulties through targeted interventions is thus crucial to promote better communication and relational outcomes for children with NDD.

The parent-child relationship serves as the primary context in which the child develops cognitive, linguistic, and social-emotional skills through contingent and synchronous interactions with the parent. However, contingent interactions between parents and children can be challenging when the child has a NDD, as their communicative behaviors may be unclear or difficult to interpret. Reduced or partial signals, such as facial expressions, gestures like pointing, reaching, or showing objects, can hinder the parents' ability to accurately interpret the child's cues and intentions, complicating the interaction and making it more difficult for parents to respond appropriately. Indeed, Indeed, alterations in early preverbal intersubjective and socio-communicative skills-such as vocalizations, eye contact, smiling, and shared attention-can disrupt the quality of daily parent-child interactions. These disruptions may negatively impact on parenting behavior, potentially leading to long-term adverse effects on the child's cognitive and language development. Involving parents in early interventions may help them perceive and understand early communicative signals of their children, enabling an appropriate response and providing suitable and contingent stimulations.

Primary aim of the study: The main aim is to compare the feasibility and efficacy of an intervention focused on socio-communicative intersubjective skills, actively involving one of the parents (SPEAK intervention), with those of standard speech therapy. The goal is to determine whether the intervention tailored to these specific skills and involving parents provides greater benefits in supporting early communication and social development.

Secondary aims of the study: A secondary aim is to evaluate whether the SPEAK intervention actively involving parents will lead to improvements in how parents interact with their children.

Exploratory aims: Additional exploratory aims of this study include: (a) verifying whether the SPEAK intervention may also result in improvements in children's socio-cognitive skills and socio-emotional development; (b) investigating associations between parenting behaviour and other outcome measures at T0 across groups; (c) assessing the psychometric properties of the recently developed tool "Observation of Prelinguistic Intersubjective and Socio-Communicative Skills" (OPISCoS; Strazzer et al., 2023), through comparisons with standardized tests that evaluate communication and social development.

Procedure: Sixty children with NDD, aged between 6 months and 5 years, will be recruited from rehabilitation centers affiliated with Associazione La Nostra Famiglia. All centers treat similar clinical populations and utilize a consistent rehabilitative approach. Eligible participants will be referred by the attending physician to the research team. Parents will be informed about the study's procedures and asked to provide informed consent.

Participants will be randomly assigned to either the experimental group, which will receive an intervention focused on socio-communicative and intersubjective skills (SPEAK intervention), or the control group, which will receive standard speech therapy (care as usual). Stratified randomization with permuted blocks will be used to ensure balanced group assignment based on age and developmental quotient. Age will be split as follows: 6 - 35 months, 36 - 59 months. The cut-off for developmental quotient will distinguish participants with moderate/severe psychomotor delay (< 55 or non-assessable) and with mild psychomotor delay/borderline functioning (≥ 55). This way, participants will be assigned to the two arms according to the permuted sequences within the four stratification blocks (16 patients per block).

Participants assigned to the experimental arm will receive eight sessions of an intervention focused on early socio-communicative and intersubjective skills, which will actively involve one of the parents. Participants assigned to the control group will receive standard speech therapy. Both interventions will be carried out by previously formed speech therapists, and will have the same duration - 8 45-minute weekly sessions, over two months.

Before starting any intervention sessions, participants will be administered with standardized tests to assess primary and secondary outcomes. Information regarding previous or concurrent rehabilitative treatments (e.g., psychomotricity), as well as other pertinent clinical and socio-demographic data (e.g., socio-economic status), will be collected from medical records or through specific questionnaires.

Adherence to the study Given the rehabilitative nature of the interventions and the fact that parents request access to rehabilitation centers for speech therapy, significant adherence challenges are not anticipated. In line with previous early intervention studies, a drop-out rate of 10-15% is expected among recruited patients. At the time of recruitment, it will be required that at least one parent attends all sessions to minimize differences in drop-out rates between the experimental and control groups, since only the experimental intervention involves active parental participation. Adherence will be monitored by recording the number of participants who discontinue treatment, documenting reasons for withdrawal where possible, and tracking the number of sessions completed by each participant.

Evaluation of the potential benefit/risk ratio for the population. No risks are anticipated for the study population. The assessments and procedures to be implemented are consistent with the activities already conducted in the clinical practice at the recruiting rehabilitation centers. The assessments conducted both at the beginning and end of intervention directly benefit participants by providing a comprehensive evaluation of their progress. Indirectly, the study will encourage a more focused approach to socio-communicative and intersubjective skills in speech therapy with children with NDD. Additionally, the study will promote the specialized training of the speech therapists involved, further enhancing care quality.

ELIGIBILITY:
Inclusion criteria:

For children:

* Age between 6 months (corrected age in cases of prematurity) and 5 years.
* Documented developmental delay and/or socio-communicative difficulties, based on clinical signs or standardized developmental scales (e.g., Griffiths Scales).
* Mental age of at least 6 months.
* Diagnosis of neurodevelopmental disability, including cerebral palsy, genetic syndromes, rare diseases with non-progressive neurological impairments, or congenital disorders of undetermined nature.

For parents:

* Adult age (≥ 18 yo)
* Good knowledge and fluency in Italian.
* No manifest psychiatric conditions.
* No documented intellectual disability.

Exclusion criteria:

For children:

* Age greater than 5 years at the time of recruitment.
* Mental age below 6 months.
* Absence of developmental delay (developmental quotient > 85) and socio-communicative difficulties.
* Diagnosis of neurodevelopmental disability resulting from neurodegenerative diseases or brain tumor outcomes.
* Severe sensory impairments (profound deafness and/or blindness).

For Parents:

* Inability to speak Italian.
* Documented psychiatric conditions or intellectual disability.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Early socio-communicative skills | Primary outcomes will be assessed at two time points: before the interventions (T0) and at the conclusion of the interventions, which will occur two months after the first session (T2).
  - Prelinguistic intersubjective and socio-communicative skills will be assessed through the observative checklist "Observation of Prelinguistic Intersubjective and Socio-Communicative Skills" (OPISCoS). The total raw score will be obtained by summing raw scores of all items. Higher scores indicate better early socio-communicative skills.
Communication and language development | Primary outcomes will be assessed at two time points: before the interventions (T0) and at the conclusion of the interventions, which will occur two months after the first session (T2).
  The MacArthur-Bates Communicative Development Inventory - short form will be fulfilled by parents to obtain an index of child language development. Higher scores indicate better developmental outcomes.
Parenting behavior | The parent-child interactions will be recorded and then coded with PICCOLO at two time points: before the interventions (T0) and at the conclusion of the interventions, which will occur two months after the first session (T2).
  A ten-minute parent-child interaction will be recorded and subsequently coded using the the "Parenting Interactions with Children Checklist of Observations Linked to Outcomes" (PICCOLO). This coding system an observational measure of developmentally supportive parental behavior, divided into four domains: affection, responsiveness, encouragement, teaching. Higher scores indicate more positive parenting behaviors.

SECONDARY OUTCOMES:
Early socio-cognitive skills | This outcome will be assessed at two time points: before the interventions (T0) and at the conclusion of the interventions, which will occur two months after the first session (T2).
  The Early Socio-cognitive Battery (ESB) will be administered to assess socio-cognitive skills, such as social responsivity, joint attention and symbolic comprehension. Raw scores will be converted into standardized scores according to normative tables. Higher scores indicate better socio-cognitive skills.
Socio-emotional development | This outcome will be assessed at two time points: before the interventions (T0) and at the conclusion of the interventions, which will occur two months after the first session (T2).
  Socio-emotional development will be evaluated through the parent-reported questionnaire of the Bayley-3 scales. Higher scores indicate better developmental outcomes.
Feasibility outcome measures | This outcome will be assessed at the conclusion of the interventions, which will occur two months after the first session (T2)
  Feasibility will be assessed by tracking the number of dropouts, namely the number of participants who fail to complete the eight-session intervention, and the number of sessions attended per child.
Acceptability and perceived efficacy measures | This outcome will be assessed at the conclusion of the interventions, which will occur two months after the first session (T2)
  At T2, parents from both the IG and CG will complete a short questionnaire to provide subjective evaluations of the intervention's acceptability and perceived efficacy. The questionnaire will assess recommendation level and satisfaction, as well as parent's perception of their child's required effort, and the difficulties encountered in initiating and maintaining the intervention

OTHER OUTCOMES:
Socio-demographic and clinical information | This information will be collected before the intervention (T0).
  Information regarding clinical (e.g., diagnosis) and socio-demographic data (e.g., socio-economic status), will be collected from medical records or through specific questionnaires.
Child behavior | This outcome will be collected before the intervention (T0).
  The parent-report Child Behavior Checklist (CBCL) 1½-5 [57,58] will be administered to assess the presence of emotional-behavioral problems (e.g., anxiety, sleep problems) in children older than 17 months. Raw scores will be converted into T-scores according to normative tables, with higher scores indicating greater problems.
Parental depressive symptoms. | This outcome will be collected before the intervention (T0).
  Parents will be asked to fulfill the Beck Depression Inventory (BDI), which assesses the presence of depressive symptoms. Higher scores indicate increased depressive symptoms.
Parental anxiety | This outcome will be collected before the intervention (T0).
  The parent-report State-Trait Anxiety Inventory (STAI-Y) will be administered to evaluate transient and stable states of anxiety. Higher scores indicate greater levels of state and trait anxiety symptomatology .
Parental stress | This outcome will be collected before the intervention (T0).
  The Parenting Stress Index (PSI) questionnaire will be adopted to provide a measure of the overall stress experienced in parenting. Higher scores represent stronger parenting stress.

CONTACTS AND LOCATIONS:
Locations (9):
- Italy (9):
  - Associazione "La Nostra Famiglia" - Centro di Riabilitazione Ambulatoriale, Como, Como
  - Associazione "La Nostra Famiglia" - Centro di Riabilitazione Ambulatoriale e Diurno (CDC), Ponte Lambro, Como
  - Associazione "La Nostra Famiglia" - Centro di Riabilitazione Ambulatoriale, Diurno (CDC) e Residenziale, Bosisio Parini, Lecco
  - Associazione La Nostra Famiglia - IRCCS E. Medea, Bosisio Parini, Lecco
  - Associazione "La Nostra Famiglia" - Centro di Riabilitazione Ambulatoriale, Diurno (CDC) e Domiciliare, Lecco, Lecco
  - Associazione "La Nostra Famiglia"- Centro di Riabilitazione Ambulatoriale, Sesto San Giovanni, Milano
  - Associazione "La Nostra Famiglia"- Centro di Riabilitazione Ambulatoriale, Carate Brianza, Monza E Brianza
  - Associazione "La Nostra Famiglia"- Centro di Riabilitazione Ambulatoriale, Cislago, Varese
  - Associazione "La Nostra Famiglia"- Centro di Riabilitazione Ambulatoriale, Diurno (CDC), Vedano Olona, Varese

IPD SHARING:
Plan to Share IPD: Yes
Anonymized raw data will be made available through public repositories, such as ZENODO.

REFERENCES:
- [Derived] Porro C, Butti N, Sacchi D, Rigamonti R, Miccoli A, Montirosso R, Strazzer S. Speech therapy and parenting for early socio-communicative skills in young children with neurodevelopmental disabilities (SPEAK): study protocol for an Italian multicentre randomised controlled trial. BMJ Open. 2025 Nov 4;15(11):e102104. doi: 10.1136/bmjopen-2025-102104. PMID 41193214